CLINICAL TRIAL: NCT05994547
Title: Safety and Efficacy of Remimazolam Compared With Midazolam During Bronchoscopy: A Single Center, Randomized Controlled Study
Brief Title: Efficacy and Safety of Remimazolam Compared With Midazolam During Bronchoscopy:Randomised Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chungbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Bumhee Yang, MD, Associator professor M.D. PhD., Chungbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Remimazolam Vs midazolam
Record Dates: First submitted 2023-07-31; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Bronchoscopy; Remimazolam
Keywords: Remimazolam; midazolam; safety; efficacy
MeSH Terms: interventions — remimazolam; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam (Experimental): Patients aged <60 years or weighing >50 kg were randomly assigned to receive 3 mg intravenous midazolam. In contrast, those aged ≥60 years or with a body weight of <50 kg were assigned 2 mg intravenous.
  If adequate sedation was not achieved after the initial sedative administration, additional midazolam (0.5 mg) was administered at intervals of 3-4 min, at the discretion of the physician.
  Interventions: Drug: Midazolam
- Remimazolam (Active Comparator): Patients aged <60 years or weighing >50 kg were randomly assigned to receive 5 mg remimazolam. In contrast, those aged ≥60 years or with a body weight of <50 kg were assigned intravenous 3 mg remimazolam.
  If adequate sedation was not achieved after the initial sedative administration, additional remimazolam (2.5 mg) was administered at intervals of 3-4 min, at the discretion of the physician.
  Interventions: Drug: Byfavo

INTERVENTIONS:
Drug: Byfavo — For induction and maintenance of sedation
  Other Names: Remimazolam
  Arms: Remimazolam
Drug: Midazolam — For induction and maintenance of sedation
  Arms: Midazolam

SUMMARY:
Objectives: Although remimazolam is an ultra-short-acting benzodiazepine with a shorter elimination half-life and faster recovery time than midazolam, studies evaluating its safety and efficacy during bronchoscopy are limited. This study compared the safety and efficacy of remimazolam with that of midazolam for bronchoscopy.

Design: A single-center, prospective randomized parallel-group study

Setting: Chungbuk National University Hospital, April 2022-June 2023.

Participants: One hundred patients were enrolled; 51 were randomly assigned to the midazolam group and 49 to the remimazolam group. Respiratory nurse specialists performed the randomization.

Interventions: Oral and laryngeal anesthesia was induced using a 4% lidocaine nebulizer prior to sedation. The vocal cords and lower airway tract were anesthetized.

Patients aged <60 years or weighing >50 kg received 3 mg intravenous midazolam or 5 mg remimazolam. Patients aged ≥60 years or weighing <50 kg received 2 mg intravenous midazolam or 3 mg remimazolam. Bronchoscopy was performed under adequate sedation (MOAA/S≤3)

Main outcome measures: The primary outcome was the time from the end of the procedure to full alertness. Secondary outcomes were procedural time parameters, satisfaction profiles, and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years who required diagnostic or therapeutic bronchoscopy and agreed to participate

Exclusion Criteria:

* 1) pregnancy, 2) moderate-to-severe hepatic impairment and lactose intolerance 3) mechanical ventilation 4) history of tracheostomy 5) poor patient cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
the time from the end of the procedure to full alertness in both groups. | up to 2 hours (MOAA/S had recovered to 5 after the procedure had been completed.)
  The Time for patient to recover Modified Observer's Assessment of Alertness and Sedation (MOAA/S) scores to 5 after end of bronchoscopy
  MOAA/S scores: 5 = Responds readily to name spoken in normal tone [alert], 4 =Lethargic response to name spoken in normal tone, 3 = Responds only after name is called loudly and/or repeatedly, 2 = Responds only after mild prodding or shaking, 1 = Responds only after painful trapezius squeeze, 0 = Does not respond to painful trapezius squeeze.
  MOAA/S scores were assessed by the investigators.
the time taken to reach peak sedation | up to 30 minutes (the time to the start of the procedure after the administration of the first dose of medication)
  The degree of sedation was measured using the Modified Observer's Alertness/Sedation scale (MOAA/S), and bronchoscopy was performed under adequate sedation (MOAA/S≤3)

SECONDARY OUTCOMES:
physician satisfaction after the procedure | up to 1day
  Physician satisfaction with sedation was expressed as a score ranging from -5 to 5 after completion of the procedure (-5 = not satisfied at all, 5 = maximally satisfied).
patient satisfaction after the procedure | up to 1day
  Patient satisfaction was measured using a visual analog scale (0 = intolerable, 10 = free from inconvenience).
difference between the adverse effects that occurred after bronchoscopy in the midazolam and remimazolam groups. | up to 30days (the first dose to the end of the procedure was defined as the time from the first sedative drug administration to mouth exit.)
  adverse effects that occur during and after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, North Chungcheong, South Korea

REFERENCES:
- [Derived] Kim SH, Cho JY, Kim M, Chung JM, Yang J, Seong C, Kim EG, Seok JW, Shin YM, Lee KM, Choe KH, Han JH, Yang B. Safety and efficacy of remimazolam compared with midazolam during bronchoscopy: a single-center, randomized controlled study. Sci Rep. 2023 Nov 22;13(1):20498. doi: 10.1038/s41598-023-47271-w. PMID 37993525